CLINICAL TRIAL: NCT04370301
Title: Pilot Study of JAK Inhibitor Therapy Followed by Reduced Intensity Haploidentical Transplantation for Patients With Myelofibrosis
Brief Title: Reduced Intensity Haploidentical Transplantation for the Treatment of Primary or Secondary Myelofibrosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1006957; NCI-2020-02422 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10441 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Primary Myelofibrosis; Secondary Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — Cyclophosphamide; Janus Kinase Inhibitors; ruxolitinib; fedratinib; fludarabine; pegylated granulocyte colony-stimulating factor; Melphalan; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Tacrolimus; Whole-Body Irradiation; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort I (JAK inhibitor, conditioning, GVHD prophylaxis) (Experimental): JAK INHIBITOR THERAPY: Patients receive a JAK inhibitor at least 8 weeks prior to the start of HCT conditioning through day -4 before transplantation.
  CONDITIONING: Patients receive melphalan IV over 1 hour on day -5, fludarabine IV over 30-60 minutes on days -5 to -2, and undergo TBI on day -1 or day -1 and day 0.
  TRANSPLANT: Patients receive peripheral blood stem cell infusion on day 0.
  GVHD PROPHYLAXIS: Patients then receive cyclophosphamide IV over 3 hours on days 3-4, tacrolimus IV beginning day 5 then PO for about 6 months, mycophenolate mofetil PO BID or TID beginning day 5 for 6 weeks, and G-CSF SC beginning day 7 until neutrophil recovery is > 1,500/mm^3.
  All patients undergo MRI, CT, bone marrow biopsy and aspiration and blood sample collection throughout the trial. Patients also undergo ECHO or MUGA on the trial.
  Interventions: Drug: Cyclophosphamide; Drug: JAK Inhibitor; Drug: Fludarabine; Biological: Recombinant Granulocyte Colony-Stimulating Factor; Drug: Melphalan; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Tacrolimus; Radiation: Total-Body Irradiation; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Bone Marrow Biopsy; Procedure: Bone Marrow Aspiration; Procedure: Biospecimen Collection; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan
- Cohort II (JAK inhibitor, conditioning, GVHD prophylaxis) (Experimental): JAK INHIBITOR THERAPY: Patients receive a JAK inhibitor at least 8 weeks prior to the start of HCT conditioning through day -4 before transplantation. Additionally, patients receive a JAK inhibitor following transplantation beginning day 5 through 9-12 months after transplant.
  CONDITIONING: Patients receive melphalan IV over 1 hour on day -5, fludarabine IV over 30-60 minutes on days -5 to -2, and undergo TBI on day -1 or day -1 and day 0.
  TRANSPLANT: Patients receive peripheral blood stem cell infusion on day 0.
  GVHD PROPHYLAXIS: Patients then receive cyclophosphamide IV over 3 hours on days 3-4, tacrolimus IV beginning day 5 then PO for about 6 months, mycophenolate mofetil PO BID or TID beginning day 5 for 6 weeks, and G-CSF SC beginning day 7 until neutrophil recovery is > 1,500/mm^3.
  All patients undergo MRI, CT, bone marrow biopsy and aspiration and blood sample collection throughout the trial. Patients also undergo ECHO or MUGA on the trial.
  Interventions: Drug: Cyclophosphamide; Drug: JAK Inhibitor; Drug: Fludarabine; Biological: Recombinant Granulocyte Colony-Stimulating Factor; Drug: Melphalan; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Tacrolimus; Radiation: Total-Body Irradiation; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Bone Marrow Biopsy; Procedure: Bone Marrow Aspiration; Procedure: Biospecimen Collection; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719; Asta B 518; B-518; WR-138719
Drug: JAK Inhibitor — Given PO
  Other Names: JAK inhibitors; Janus Kinase Inhibitor; Ruxolitinib; Fedratinib
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Biological: Recombinant Granulocyte Colony-Stimulating Factor — Given SC
  Other Names: Recombinant Colony-Stimulating Factor 3; rhG-CSF; 143011-72-7
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine mustard; L-sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Procedure: Peripheral Blood Stem Cell Transplantation — Given IV
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; peripheral stem cell support; Peripheral Stem Cell Transplant; peripheral stem cell transplantation
Drug: Tacrolimus — Given IV and PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic; FK-506; Tacforius
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TBI; Total Body Irradiation; Whole Body Irradiation; Whole-Body Irradiation; Total-Body Irradiation Prior to Stem Cell Transplant; SCT_TBI
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT Scan; Computed Axial Tomography; CT SCAN
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MR Imaging; MRI
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and aspiration
  Other Names: Biopsy of Bone Marrow
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and aspiration
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning

SUMMARY:
This initial cohort of this phase II trial studied the outcomes of using a JAK inhibitor prior to reduced intensity haploidentical (Haplo) transplantation for the treatment of primary or secondary myelofibrosis (MF). The primary risk of using Haplo HCT in patients with MF is graft failure. In the first cohort, all patients engrafted. There were no instances of graft failure. However, a large number of patients did have graft versus host disease as a complication of their transplant. JAK inhibitors have since been approved for the indication of graft versus host disease treatment. And we are also using them for graft versus host disease prevention in a study of MF patients with sibling and unrelated donors. Therefore, we are opening a new cohort of the current study using the JAK inhibitor prior to, during and after Haplo transplant. Our goal is to decrease graft versus host disease in patients receiving a Haplo MF transplant without increasing the risk of graft failure.

DETAILED DESCRIPTION:
OUTLINE: Cohort 1 is now closed and all patients will be enrolled on Cohort 2.

COHORT I:

JAK INHIBITOR THERAPY: Patients receive a JAK inhibitor at least 8 weeks prior to the start of hematopoietic cell transplantation (HCT) conditioning through day -4 before transplantation.

CONDITIONING: Patients receive melphalan intravenously (IV) over 1 hour on day -5, fludarabine IV over 30-60 minutes on days -5 to -2, and undergo total-body irradiation (TBI) on day -1 or day -1 and day 0.

TRANSPLANT: Patients receive peripheral blood stem cell infusion on day 0.

GVHD PROPHYLAXIS: Patients then receive cyclophosphamide IV over 3 hours on days 3-4, tacrolimus IV beginning day 5 then orally (PO) for about 6 months, mycophenolate mofetil PO twice daily (BID) or three times daily (TID) beginning day 5 for 6 weeks, and granulocyte colony-stimulating factor (G-CSF) subcutaneously (SC) beginning day 7 until neutrophil recovery is > 1,500/mm^3.

COHORT II:

JAK INHIBITOR THERAPY: Patients receive a JAK inhibitor at least 8 weeks prior to the start of HCT conditioning through day -4 before transplantation. Additionally, patients receive a JAK inhibitor following transplantation beginning day +5 through 9-12 months after transplant.

CONDITIONING: Patients receive melphalan IV over 1 hour on day -5, fludarabine IV over 30-60 minutes on days -5 to -2, and undergo TBI on day -1 or day -1 and day 0.

TRANSPLANT: Patients receive peripheral blood stem cell infusion on day 0.

GVHD PROPHYLAXIS: Patients then receive cyclophosphamide IV over 3 hours on days 3-4, tacrolimus IV beginning day 5 then PO for about 6 months, mycophenolate mofetil PO BID or TID beginning day 5 for 6 weeks, and G-CSF SC beginning day 7 until neutrophil recovery is > 1,500/mm^3.

All patients undergo magnetic resonance imaging (MRI), computed tomography (CT), bone marrow biopsy and aspiration and blood sample collection throughout the trial. Patients also undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) on the trial.

After completion of study treatment, patients are followed up between day 80-100, at 1 year, and then up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* PART 1: JAK INHIBITOR ADMINISTRATION INCLUSION CRITERIA
* Age between 18 and 70 years
* Diagnosis of primary myelofibrosis (PMF) as defined by the 2016 World Health Organization classification system or diagnosis of secondary MF as defined by the International Working Group (IWG) for Myeloproliferative Neoplasms Research and Treatment criteria
* Patients meeting the criteria for intermediate-1, intermediate-2 or high-risk disease by the Dynamic International Prognostic Scoring System (DIPSS)-plus scoring system (DIPSS may be used if all data from DIPSS are not available)
* Ability to understand and the willingness to sign a written informed consent document (or legally authorized representative)
* Patient must be a potential hematopoietic stem cell transplant candidate
* PART 2: ALLOGENEIC STEM CELL TRANSPLANT INCLUSION CRITERIA
* Meeting criteria for 1st phase as above, at time of initiation of JAK inhibitor, including ability to understand and willingness to sign a written informed consent (or legally authorized representative). Patients arriving to our institution for transplant and not enrolled in Part 1 may still be enrolled in Part 2 if Part 1 criteria met. These patients will have Part 1 endpoints transcribed from medical records
* Received JAK inhibitor for at least 8 weeks immediately prior to conditioning and be willing to continue until 9-12 months post-transplant as tolerated
* Karnofsky performance status score >= 70
* Calculated creatinine clearance using the Cockcroft-Gault formula or 24 hour (hr) urine creatinine clearance must be > 60 ml/min
* Total serum bilirubin must be < 3 mg/dL unless the elevation is thought to be due to Gilbert's disease or hemolysis
* Transaminases must be < 3 x the upper limit of normal
* Patients with clinical or laboratory evidence of liver disease will be evaluated for the cause of liver disease, its clinical severity in terms of liver function, and the degree of portal hypertension. Patients with fulminant liver failure, cirrhosis with evidence of portal hypertension or bridging fibrosis, alcoholic hepatitis, hepatic encephalopathy, or correctable hepatic synthetic dysfunction evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, and symptomatic biliary disease will be excluded
* Diffusion capacity of the lung for carbon monoxide (DLCO) corrected > 60% normal; may not be on supplemental oxygen
* Left ventricular ejection fraction > 40% OR shortening fraction > 26%
* Comorbidity Index < 5 at the time of pre-transplant evaluation
* DONOR: Patients must be screened prior to transplant for donor-specific anti-HLA antibodies (DSA). Patients with DSA will be reviewed by the principal investigator and considered for desensitization treatment
* DONOR: Children are preferred over siblings and parents
* DONOR: Younger donors are preferred over older donors
* DONOR: ABO matched donors are preferred over minor ABO mismatched and over major ABO mismatch donors

Exclusion Criteria:

* PART 1: JAK INHIBITOR ADMINISTRATION EXCLUSION CRITERIA
* Contraindication to receiving a JAK inhibitor including:

  * Patients who have known hypersensitivity to JAK inhibitors
  * Clinical or laboratory evidence of significant renal or hepatic impairment including cirrhosis
  * Active uncontrolled infection
  * Known human immunodeficiency virus (HIV) positivity
  * Women who are pregnant or trying to conceive
  * Caution should be used in patients with platelets < 100 though adjustments in dose can be made to accommodate anyone with platelets > 50
* History of prior allogeneic transplant
* Leukemic transformation (> 20% blasts)
* PART 2: ALLOGENEIC STEM CELL TRANSPLANT EXCLUSION CRITERIA
* Uncontrolled viral or bacterial infection at the time of study enrollment
* Active or recent (prior 6 month) invasive fungal infection without infectious disease (ID) consult and approval
* Known HIV positivity
* Pregnant or breastfeeding
* Availability of an human leukocyte antigen (HLA)-identical or 1-allele-mismatched related donor or an HLA 10 of 10 matched unrelated donor

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Probability of primary and secondary graft failure | Up to 5 years
  Primary graft failure is defined as failure to achieve an absolute neutrophil count of > 500/ul by 42 days after bone marrow or peripheral blood stem cell transplantation. Secondary graft failure is defined as cytopenias after initial engraftment, with (a) donor chimerism of < 5% or (b) falling donor chimerism with intervention such as second transplant or donor lymphocyte infusion or (c) patient death due to cytopenias, and fall in donor chimerism, even if chimerism is > 5%. Exclusion criteria for diagnosis of graft failure are (a) disease relapse, (b) graft-versus-host disease, and (c) other causes of cytopenias such as, viral infection and drug toxicity.

SECONDARY OUTCOMES:
Incidence of severe (grade 3 or 4) cytokine release syndrome | Up to 5 years
Non-relapse mortality (NRM) | Day 100
NRM | 1 year
Overall survival | 1 year
Overall survival | 3 years
Incidence of grade II-IV acute graft versus host disease (GVHD) | Up to 5 years
Incidence of grade III-IV acute GVHD | Up to 5 years
Incidence of moderate-severe chronic GVHD | Up to 5 years
Incidence of relapse | At 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rachel B. Salit, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No